CLINICAL TRIAL: NCT06439979
Title: Rural Adult and Youth Sun Protection Study - Rural Baseball R01
Brief Title: Rural Adult and Youth Sun Protection Study
Acronym: RAYS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Georgetown University (Other); West Virginia University (Other)
Responsible Party: Principal Investigator, Yelena Wu, Associate Professor, Department of Dermatology; Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00173007
Record Dates: First submitted 2024-05-13; First posted 2024-06-03 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Melanoma (Skin); Skin Cancer
Keywords: Rural; Melanoma, Skin cancer; Prevention; Underserved communities; Youth; Sports
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: RAYS uses a 2-arm cluster-randomized trial in 2 rural US states (Utah and West Virginia) matched for high skin cancer burden and rurality. This parallel model includes an intervention arm, which will include sun-safety education and skin cancer prevention, and the control arm which will focus on general sports-related injury prevention. Leagues enrolled in the study will be randomized to one of the two arms.
Who Masked: Participant
Masking Description: Masking will only be used for participants in the study. Investigators will know which arm of the study each participant has been randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAYS Intervention (Experimental): The RAYS arm is the intervention being tested, which will include skin cancer prevention education and providing participants with sun-safety supplies.
  Interventions: Behavioral: RAYS Intervention
- Control (No Intervention): The Control arm of the study will not receive any skin cancer prevention information or sun-safety materials but will only receive general injury prevention information.

INTERVENTIONS:
Behavioral: RAYS Intervention — Developmental baseball leagues will be randomly assigned to RAYS vs. control. Outcomes include directly-observed child sun safety behaviors after controlling for environmental ultra-violet radiation (UVR), with parent-reported child sun protection and other related endpoints at 1 year.
  Arms: RAYS Intervention

SUMMARY:
The purpose of this study is to help prevent skin cancer by improving the use of sun protective behaviors among youths living in rural communities in Utah and West Virginia.

DETAILED DESCRIPTION:
Children living in rural and under-served communities are at high risk for skin cancer; however, there are no evidence-based sun safety interventions showing durable effects for this vulnerable pediatric population. The objective of this proposal is to rigorously test a novel, multi-level approach to skin cancer prevention among young rural children that is delivered through developmental baseball leagues. To attain this objective, the investigators will conduct a two-arm cluster-randomized trial with the primary outcome being multi-behavior sun protection change among children.

ELIGIBILITY:
Parent inclusion criteria:

i. Adults who currently have children ages 3 and older years of age playing on participating sports teams in leagues serving rural areas in Utah or West Virginia (rural is defined as ≥4 by the RUCA or RUCC systems)

ii. Live and/or work in rural communities in Utah or West Virginia (≥4 as defined by the RUCA or RUCC systems)

Coach/leader inclusion criteria:

i. Adults who serve as coaches or leaders of recreational sports (i.e. baseball/softball, soccer, flag football, etc.) teams or developmental programs serving children ages 3 and older

ii. Live and/or work in rural areas of Utah or West Virginia (rural is defined as ≥4 by the RUCA or RUCC systems)

Participant inclusion criteria for minor participants (ages 3 and older) are as follows:

i. Live in rural communities and/or participate in sports leagues serving rural communities in Utah or West Virginia (≥4 as defined by the RUCA or RUCC systems).

Participant inclusion criteria for key informant interviews are as follows:

i. Adults who serve as leaders or who are affiliated with sports leagues or community groups serving rural youths and/or adults who currently have minor children 3 years of age or older playing on participating sports teams and/or adults who live and/or work in rural communities in Utah or West Virginia ((≥4 as defined by the RUCA or RUCC systems)

Local sports leagues will be eligible to participate if they convene recreational sports (i.e. baseball/softball) teams or developmental programs (i.e. T-ball and coach pitch) for children ages 3 and older.

Exclusion Criteria:

* Adults and children who do not speak or read English will be excluded.
* For individuals asked to complete surveys, individuals who have a medical or other condition (e.g., developmental delay) that would preclude their completion of these surveys will be excluded.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 843 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Directly observed child sunscreen application | At baseline and post-intervention (3-6 weeks after intervention has been delivered)
  Teams and their players will be observed once at the beginning and once at the end of the baseball season. A trained research assistant will tally the total number of children who applied sunscreen at any time during the practice or game. This tallied number will create a percentage of the team that applied sunscreen. The percentages from the beginning and end of the season will be compared to determine the effectiveness of the intervention.
  "How many wearing sunscreen?" Higher percentages indicate higher proportion of players on the team who engaged in that sun protective behavior.
Directly observed child hat wearing | At baseline and post-intervention (3-6 weeks after intervention has been delivered)
  Teams and their players will be observed once at the beginning and once at the end of the baseball season. A trained research assistant will tally the total number of children who wore a hat at any time during the practice or game. This tallied number will create a percentage of the team that wore a hat. The percentages from the beginning and end of the season will be compared to determine the effectiveness of the intervention.
  "How many wore a hat?" Higher percentages indicate higher proportion of players on the team who engaged in that sun protective behavior.
Directly observed child wearing long sleeves | At baseline and post-intervention (3-6 weeks after intervention has been delivered)
  Teams and their players will be observed once at the beginning and once at the end of the baseball season. A trained research assistant will tally the total number of children who wore a long-sleeved shirt at any time during the practice or game. This tallied number will create a percentage of the team that wore protective long-sleeved shirts. The percentages from the beginning and end of the season will be compared to determine the effectiveness of the intervention.
  "How many wore long sleeves?" Higher percentages indicate higher proportion of players on the team who engaged in that sun protective behavior.
Directly observed child shade seeking | At baseline and post-intervention (3-6 weeks after intervention has been delivered)
  Teams and their players will be observed once at the beginning and once at the end of the baseball season. A trained research assistant will tally the total number of children who spent time in shade or under an umbrella at any time during the practice or game. This tallied number will create a percentage of the team that spent time in shade/under umbrella. The percentages from the beginning and end of the season will be compared to determine the effectiveness of the intervention.
  "How many in shade/under umbrella?" Higher percentages indicate higher proportion of players on the team who engaged in that sun protective behavior.

SECONDARY OUTCOMES:
Parent-reported child sun protection behaviors | At baseline, post-intervention (3-6 weeks after intervention has been delivered), and one year post-baseline
  A random sample of parents will report on their child's use of sun protection using the Sun Habits Survey, a well-established and valid measure. These same parents will be asked to complete questionnaires at baseline, end-of-season, and at 1 year follow-up.
  "On a warm and sunny day, how often did your child...Use sunscreen with a sun protective factor (SPF) of 30+?" All parent-reported items will be assessed on a 5-point Likert-type scale ("Never" to "Always").
Parent-report child sunburn | At baseline, post-intervention (3-6 weeks after intervention has been delivered), and one year post-baseline
  Parents will report on the number of sunburns their child experienced during baseball and not during baseball at baseline, post-intervention and one-year post-baseline. Parents will report on child behaviors using items from the Sun Habits Survey.
  "How many times did your child have a red OR painful sunburn that lasted a day or more? In the past month? In the past 12 months?" Minimum value = 0, maximum value = 5 or more.
  A low number indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yelena P Wu, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Informed Consent Form: ICF_Utah_Coaches (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT06439979/ICF_000.pdf
  • Informed Consent Form: ICF_Utah_Parents (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT06439979/ICF_001.pdf
  • Informed Consent Form: ICF_Utah_CommunityMembers (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT06439979/ICF_002.pdf